CLINICAL TRIAL: NCT00115882
Title: Proactive Smoking Cessation for Adolescents
Brief Title: Hutchinson Study of High School Smoking
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FHCRC IRB #4727; R01CA082569 (NIH)
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Smoking Cessation
Keywords: Adolescent; smoking; smoking cessation; counseling
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): proactive smoking-cessation telephone counseling
  Interventions: Behavioral: MI + CBST
- 2 (No Intervention): no-intervention control

INTERVENTIONS:
Behavioral: MI + CBST — The HS Study intervention consisted of proactive identification and recruitment of eligible smokers (and selected nonsmokers) within the target population, and a protocol-guided series of counselor-initiated, personally-tailored telephone calls (from 1 to 10, depending on participant's interest) to eligible high school senior smokers and nonsmokers in experimental high schools. The telephone-delivered behavioral intervention integrated Motivational Interviewing and Cognitive Behavioral Skills building. Content and dose were tailored to the individual.
  Other Names: HS Study Intervention
  Arms: 1

SUMMARY:
The primary goal of the Hutchinson Study of High School Smoking, a group-randomized trial conducted by the Fred Hutchinson Cancer Research Center in partnership with 50 Washington State high schools, is to develop and evaluate an innovative proactive smoking cessation intervention, based upon Motivational Interviewing (MI) and Cognitive Behavioral Skills Training (CBST), for its effectiveness in reaching teen smokers and helping them succeed in quitting smoking. A positive finding would have significant implications for reducing youth smoking and, ultimately, improving the nation's health.

DETAILED DESCRIPTION:
Rates of smoking prevalence among US adolescents remain unacceptably high, with 24% of high school seniors smoking monthly and 16% smoking daily. Unfortunately, without intervention, for the majority of these adolescent smokers, smoking will be a long-term addiction. Recent studies have demonstrated that a majority of teen smokers want to quit and try to do so, but with little success.

The Hutchinson Study of High School Smoking is a 2-arm group-randomized trial in adolescent smoking cessation, conducted by the Fred Hutchinson Cancer Research Center in partnership with 50 Washington State high schools. Twenty-five high schools are randomly assigned to the experimental (intervention) condition and 25 are assigned to the control (no intervention) condition. The trial uses innovative and rigorous trial design and methodology to address recruitment, retention, and other methodological challenges encountered in early adolescent cessation trials, to provide a rigorous test of in innovative proactive smoking cessation intervention. Participants are 2,151 high school students (all smokers and a sample of nonsmokers identified via baseline survey of all enrolled students at the end of their junior year).

The intervention, delivered during the senior year of high school, consists of a series of counselor-initiated, individually-tailored telephone counseling calls. Incorporating both Motivational Interviewing and Cognitive Behavioral skills training, the counseling telephone calls aim to increase smokers' motivation for quitting smoking, build skills for smoking cessation, and assist with relapse prevention. For nonsmokers, the telephone calls provide positive reinforcement of students' abstinence choices and help build skills for supporting peers' efforts to quit smoking. Complementary intervention components include an interactive cessation/informational Web site (www.Matchbreaker.org) and school-based promotional materials (cessation posters, school newspaper ads).

Participants are followed to two follow-up times: the first at age 19 (approximately 6 months post-high school), and the second at age 25, to assess immediately after high school, and again in young adulthood, the intervention's impact on cessation status, number of quit attempts, change in readiness to quit and reduction in frequency and level of smoking.

Concerning effectiveness in reaching teen smokers, 65.3% (691 out of 1058) smokers in the intervention condition were successfully recruited, and participated in the telephone counseling.

Concerning effectiveness in helping teen smokers quit smoking, at the first follow-up, the intervention increased the percentage who achieved 6-month prolonged smoking abstinence among all smokers (21.8% in the experimental condition vs 17.7% in the control condition, difference = 4.0%, 95% confidence interval [CI] = -0.2 to 8.1, P = .06) and in particular among daily smokers (10.1% vs 5.9%, difference = 4.1%, 95% CI = 0.8 to 7.1, P = .02). There was also generally strong evidence of intervention impact for 3-month, 1-month, and 7-day abstinence and duration since last cigarette (P = .09, .015, .01, and .03, respectively). The intervention effect was strongest among male daily smokers and among female less-than-daily smokers.

ELIGIBILITY:
Inclusion Criteria:

* All high school juniors enrolled in a participating high school who reported on their baseline survey that they smoked once a month or more; and a selected sample of nonsmoker respondents (former smokers and never smokers with close friends who smoke)
* Written or verbal parental consent required for intervention participation by students under age 18

Exclusion Criteria:

* Enrolled in participating school at time of baseline survey, but not developmentally able to independently complete the baseline survey
* Not able to understand or speak English sufficiently to complete informed consent for telephone counseling
* Foreign exchange students

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2151 (Actual)
Dates: Start 2000-09; Primary Completion 2014-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
6-months prolonged smoking abstinence at age 19 and at age 25 | 6 months

SECONDARY OUTCOMES:
smoking abstinence | 3-months, 1-month, and 7-day
number of quit attempts in past 12 months | 12 months
longest length of time without smoking in past 12 months | 12 months
reduction in frequency/level of smoking | current; last 30 days
change in readiness to quit | current
change in stage of change
composite of quit duration and number of cigarettes per day | past 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Arthur V. Peterson, Jr., PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Background] Kealey KA, Ludman EJ, Mann SL, Marek PM, Phares MM, Riggs KR, Peterson AV Jr. Overcoming barriers to recruitment and retention in adolescent smoking cessation. Nicotine Tob Res. 2007 Feb;9(2):257-70. doi: 10.1080/14622200601080315. PMID 17365757
- [Background] Liu J, Peterson AV Jr, Kealey KA, Mann SL, Bricker JB, Marek PM. Addressing challenges in adolescent smoking cessation: design and baseline characteristics of the HS Group-Randomized trial. Prev Med. 2007 Aug-Sep;45(2-3):215-25. doi: 10.1016/j.ypmed.2007.05.018. Epub 2007 Jun 4. PMID 17628650
- [Result] Kealey KA, Ludman EJ, Marek PM, Mann SL, Bricker JB, Peterson AV. Design and implementation of an effective telephone counseling intervention for adolescent smoking cessation. J Natl Cancer Inst. 2009 Oct 21;101(20):1393-405. doi: 10.1093/jnci/djp318. Epub 2009 Oct 12. PMID 19822837
- [Result] Peterson AV Jr, Kealey KA, Mann SL, Marek PM, Ludman EJ, Liu J, Bricker JB. Group-randomized trial of a proactive, personalized telephone counseling intervention for adolescent smoking cessation. J Natl Cancer Inst. 2009 Oct 21;101(20):1378-92. doi: 10.1093/jnci/djp317. Epub 2009 Oct 12. PMID 19822836
- [Derived] Peterson AV Jr, Marek PM, Kealey KA, Bricker JB, Ludman EJ, Heffner JL. Does Effectiveness of Adolescent Smoking-Cessation Intervention Endure Into Young Adulthood? 7-Year Follow-Up Results from a Group-Randomized Trial. PLoS One. 2016 Feb 1;11(2):e0146459. doi: 10.1371/journal.pone.0146459. eCollection 2016. PMID 26829013
- See also: Fred Hutchinson Cancer Research Center — http://www.fredhutch.org